CLINICAL TRIAL: NCT03485573
Title: Improvement of Trauma Care Quality by Implement Trauma Register in a Middle Income Country
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Moi Univeristy (Other)
Responsible Party: Principal Investigator, Maria Lampi, Principal Investigator, RN, PhD, University Hospital, Linkoeping
Other Study IDs: KMC-002
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every year more people die from traumatic injuries than from infections such as malaria, tuberculosis, and HIV/AIDS. About 3000 people are killed annually on Kenyan roads. Hospital trauma registers have played a key role in the advancement of patient-based research and trauma care. Trauma registers offer a unique opportunity to document patient characteristics and audit outcomes, thereby creating a platform for clinical research. One of these systems is the ICD-based Injury Severity Score (ICISS) derived from and validated on hospital data to predict hospital death. The establishment of the register enables us to compare the trauma care quality with other existing or upcoming trauma registers, in different settings.

DETAILED DESCRIPTION:
The mortality caused by traumatic injuries in Africa is 116 per 100,000 population, compared to Europe with 49/100,000 population . In Kenya, which is a middle-income country in East Africa, the mortality caused by injuries is 101/100,000 population . Injuries, particularly those sustained through road traffic accidents, are a major cause of death in the African region. Statistics from the WHO reveal that, in 2015, 26.6/100,000 died in road traffic accidents in Africa. The corresponding numbers for Europe were 9.3/100,000 population . About 3000 people are killed annually on Kenyan roads, with an estimated road fatality rate of 29.1/100,000 population the affected predominantly from a productive young adult population.

MOI University/Moi Teaching and Referral Hospital (MTRH) Eldoret, Kenya, is the second national referral hospital in Kenya with a catchment of over 22 million people. A previous study, focuses on evaluating the possible benefit of in-hospital triage for trauma patients admitted to the ED at the MTRH. The study illustrated a significant need for improvement in trauma care management and also resulted in the creation of a trauma database containing ICD codes and specific patient parameters.

Although receiving increased attention, implementing strategies to improve trauma care in developing countries to address the health burden on the emergency care service is still warranted. Improved road safety legislation, reducing drunk driving, development of pre-hospital care systems , and strengthened hospital trauma care have been suggested as interventions to mitigate this problem in the health care system .

Hospital trauma registers have played a key role in the advancement of patient-based research and trauma care. Trauma registers offer a unique opportunity to document patient characteristics and audit outcomes, thereby creating a platform for clinical research. Several scoring systems to assess injury severity with the aim of improving trauma care quality have been developed. One of these systems is the ICD-based Injury Severity Score (ICISS) derived from and validated on hospital data to predict hospital death. This powerful tool uses survival risk ratios (SRRs) to calculate the probability of survival for patients and allows accurate estimates of injury severity. To calculate ICISS, each ICD-code is assigned a SRR. Each SRR is equal to the proportion of patients who survived with a specific ICD-code in a reference population. In literature searches, there is lack of published SRRs from low income countries' trauma population.

The Institutional Research and Ethics Committee (IREC) at MOI University and MOI Teaching and Referral Hospital reviewed and approved the research proposal and has been granted a Formal Approval Number (FAN: IREC 3008).

ELIGIBILITY:
Inclusion Criteria:

Trauma patients of ages 14 and above admitted to the ED at MTRH will be included in the study.

-

Exclusion Criteria:

Those brought in dead, revisits, or referred patients will excluded.

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients of ages 14 and above admitted to the ED at MTRH will be included in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Score injury severity with the aim of improving trauma care by using the ICD-based Injury Severity Score (ICISS) derived from and validated on hospital data to predict hospital death. | two years
  To calculate ICISS, each ICD-code is assigned a survival risk ratios (SRR), which represents a true continuous variable that takes on values between 0 and 1. SRR is based on the assumption that a patient's probability of survival can be predicted based on the survival rates of prior patients with similar injuries as classified by the ICD-10.
  The ICISS value is the product of SRRs from each injury sustained. A multiplicative prediction model with an assumption that all injuries contribute to the overall severity. The SRR for each code is empirically derived from the upcoming patient data. To obtain ICISS, SRRs of all injuries are multiplied.
  ICISS = SRRinj1 × SRRinj2 × SRRinj3 × SRRinj4. Create a ICISS trauma registry is valuable to document epidemiology, process and outcome, thus enabling the measurement of the impact of trauma care following injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Moi Teaching and Referral Hospital, Kenya., Eldoret, Kenya